CLINICAL TRIAL: NCT01961219
Title: Manipulation Under Anesthesia Versus Arthroscopic Capsular Release in the Treatment of Adhesive Capsulitis: A Comparison.
Brief Title: Manipulation Under Anesthesia Versus Arthroscopic Capsular Release in the Treatment of Adhesive Capsulitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficent enrollment
Sponsor: Akin Cil (Other)
Responsible Party: Sponsor-Investigator, Akin Cil, M.D., University of Missouri, Kansas City
Organization: University of Missouri, Kansas City (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-775
Record Dates: First submitted 2013-10-04; First posted 2013-10-11 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Adhesive Capsulitis of the Shoulder
MeSH Terms: conditions — Bursitis | interventions — Joint Capsule Release

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adhesive Capsulitis with MUA (Active Comparator): Subjects with idiopathic adhesive capsulitis in the "frozen" or "thawing" phase who have failed pain management and failed improvement in range of motion after at least 3 months of supervised, regimented conservative treatment; or who after less than 3 months of conservative treatment demand a quicker return to function. Treatment closed manipulation under anesthesia.
  Interventions: Procedure: Manipulation Under Anesthesia
- Adhesive Capsulitis with Arthroscopy (Active Comparator): Subjects with idiopathic adhesive capsulitis in the "frozen" or "thawing" phase who have failed pain management and failed improvement in range of motion after at least 3 months of supervised, regimented conservative treatment; or who after less than 3 months of conservative treatment demand a quicker return to function. Treatment Arthroscopic Capsular Release
  Interventions: Procedure: Arthroscopic capsular release

INTERVENTIONS:
Procedure: Manipulation Under Anesthesia — Closed manipulation under anesthesia.
  Other Names: MUA
  Arms: Adhesive Capsulitis with MUA
Procedure: Arthroscopic capsular release — Arthroscopic capsular release
  Arms: Adhesive Capsulitis with Arthroscopy

SUMMARY:
Shoulder pain is one of the most common causes of musculoskeletal disability in the adult population. Adhesive capsulitis is one of a multitude of reasons that can cause shoulder pain and dysfunction. It is a painful and disabling condition that can cause frustration for patients and caregivers due to slow recovery time. It is important to meticulously diagnose the source of the symptoms. Adhesive capsulitis is treatment by non-operative therapies such as physical therapy, exercise, steroids & pain medications. For some patients a quicker return to function is necessary; in th is situation an operative treatment is an option. This study will compare two surgical techniques for adhesive capsulitis.

Purpose

1. To directly compare outcomes of patients with adhesive capsulitis who have failed pain management and failed improvement in range of motion after at least 3 months of supervised, regimented conservative treatment and have subsequently been randomized to either closed manipulation under anesthesia or arthroscopic capsular release.
2. To blind both patient and assessing physician/nurse study coordinator to the treatment that was received for the duration of the study. This will reduce the effect of any potential bias on the results as much as possible.
3. To collect outcome data, both subjectively from the patient using proven outcome measures, and objectively from regularly spaced follow up visits with blinded assessors.
4. To collect and comment on data from the two treatment groups regarding duration of post-operative narcotic use, duration of post-operative physical therapy required, post-operative pain levels, and elapsed time until back to work/activity post-operatively.

DETAILED DESCRIPTION:
Shoulder pain is one of the most common causes of musculoskeletal disability in the adult population. Adhesive capsulitis is one of a multitude of pathologic entities that can cause shoulder pain and dysfunction. The condition is seen frequently in the clinics of primary care providers and orthopedic surgeons. Patients who develop adhesive capsulitis will typically present with complaints of pain and a progressive loss of active and passive motion of the shoulder.

The disease course of adhesive capsulitis has been extensively studied. Despite this, controversy remains as to the natural history of the disease. It is generally believed that adhesive capsulitis is a self-limiting process typically lasting twelve to thirty-six months. In one retrospective study of 50 patients with 10 year follow up, Miller et al7 found significant improvement in range of motion and resolution of pain in all patients treated conservatively. In another study, it was shown that 90% of patients treated with a stretching exercise program alone reported satisfactory outcomes at a mean follow up of 22 months8. This would mean that up to 10% of patients suffer from long-term problems. Shaffer et al9, however, reported that 50% of patients treated nonoperatively still complained of some residual pain, stiffness, or both at an average follow up of 7 years. Despite evidence that the disease improves without any intervention, many patients do not want to wait potentially as long as two to three years for resolution. For these patients, it is not unreasonable to proceed with interventions aimed at resolution of pain and improvement of motion. Levine et al10 provided some insight into predicting which patients might benefit most from proceeding with surgery. He found that patients who report more severe symptoms, are younger in age at symptom onset, and continue to have a reduction in motion after at least four months of physical therapy were more likely to eventually require surgery.

The course of progression of untreated adhesive capsulitis is described as a continuum of three clinical phases4. The first phase is characterized by pain and is termed the 'freezing' phase. In this phase, patients experience a gradual onset of diffuse shoulder pain that is progressive over a course of weeks to months. In general, pain will begin before any restriction of motion. Patients may report pain at night and often relate difficulty sleeping on the affected side. As use of the arm decreases secondary to pain, stiffness begins to set in. Phase two is characterized by stiffness and is known as the 'frozen' phase. This phase may last four to twelve months. Patients will see their pain slowly decrease, however, the limitation in motion continually increases. Phase three is known as the 'thawing' phase and may last from five to twenty-six months. This is characterized by resolution of pain and slow improvement in range of motion. Most authors agree that a longer 'freezing' phase is associated with a longer 'thawing' phase.

Adhesive capsulitis is initially treated with nonoperative therapies. The goals of conservative management are control of pain and improvement or maintenance of range of motion. Nonsteroidal anti-inflammatory medications may be prescribed to help control pain. Physical therapy with or without a home exercise program is always employed. This should be done in a gentle manner and without causing too much pain. Treatment with oral or injectable corticosteroids makes theoretical sense given the proven inflammatory nature of the condition. Studies examining treatment with oral steroids versus placebo or no treatment have yielded only short-term improvement of a few weeks. No improvement has been shown at long-term follow up of six to eight months1. There have also been many studies examining the role of intra-articular steroid injections in the treatment of adhesive capsulitis. Similarly, these studies have also shown short term (3weeks) improvement in pain and function but this improvement does not hold up at longer follow up (3-6 months)1. Jones et al11 looked at the role of suprascapular nerve blocks as a treatment option and found significant improvement in pain and shoulder range of motion at three months follow up compared to the group of patients receiving an intra-articular injection of corticosteroid. This suggests a benefit in the short-term but there is no long-term data to reveal if this improvement is lasting. Limited investigation has been performed to determine a role for hydrodilation as a viable treatment option. This involves injection of enough fluid intra-articularly to cause capsular rupture. No level I studies have been performed and only one level II study has been done which suggests some improvement in pain and Constant score up to six months1. Closed Manipulation Under Anesthesia (MUA) has been tested in short and long-term follow up and is proven to be a beneficial tool in the treatment of adhesive capsulitis in patients who have failed other nonoperative therapies. In a report on the results of MUA performed for patients with stage 2 adhesive capsulitis, Dodenhoff et al12 reported that 94% were satisfied with the procedure at mean follow up of 11 months. In a look at long-term outcomes of MUA, Farrell et al13 showed improvement in pain and motion that was continued at an average of 15 year follow up via patient questionnaire. There has been a recent trend toward arthroscopic capsular release in the treatment of refractory adhesive capsulitis and this treatment option has now become more popular than MUA. This rise in popularity of arthroscopic capsular release has occurred because of the perceived benefits of improved outcome and lower risk of complications even though there have not been any higher level trials comparing the two options. Ogilvie-Harris et al14, in a level III study, reported on a cohort of his patients treated with arthroscopic capsular release. He noted that his patients were twice as likely to be pain free at 2 year follow up as a similar cohort who underwent manipulation under anesthesia. Pollock et al15 reported in a level IV study, 83% excellent or satisfactory results after arthroscopic debridement of the rotator interval had been performed concomitantly with MUA. Warner et al16 was able to demonstrate significant improvement in all of his patients treated with arthroscopic capsular release who had failed MUA. This level IV study was performed on patients being treated for postoperative shoulder stiffness, however; not adhesive capsulitis. Both surgical methods (MUA and arthroscopic capsular release are used in our practice.

ELIGIBILITY:
Inclusion Criteria:

* patients must be diagnosed as having idiopathic adhesive capsulitis in the 'frozen' or 'thawing' phase of disease and have tried and failed at least 3 months of nonoperative therapy.

OR

* patient with adhesive capsulitis who presents already in the 'frozen' or 'thawing' phase who demands a quicker return to function and will not try 3 months of nonoperative therapy first.
* Age 18 or older

Exclusion Criteria:

* pregnancy
* previously operated shoulder (same side)
* other documented source of shoulder pain and stiffness (same side)
* rotator cuff tear (same side)
* glenohumeral osteoarthritis (same side)
* calcific tendonitis (same side)
* impingement (same side)
* osteonecrosis
* neoplasm
* cervical radiculopathy
* patients who are medically unfit to undergo a general anesthetic
* patients who are unable to comply with the post-operative protocol
* non-English Speaking patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
quick Disabilities of the arm, shoulder, and hand (quickDASH) score. | 12 months post-operatively
  The primary analysis will compare the quickDASH score at the twelve month evaluation between closed manipulation under anesthesia and arthroscopic capsular release using analysis of covariance using the baseline assessment of quickDASH ast he covariate

SECONDARY OUTCOMES:
quickDASH score | 2 weeks post-operatively
  Secondary analysis will look at all longitudinal evaluation time points of quickDASH using a mixed linear regression model to account for correlations across subjects at multiple time points.
quickDASH score | 4 weeks post-operatively
  Secondary analysis will look at all longitudinal evaluation time points of quickDASH using a mixed linear regression model to account for correlations across subjects at multiple time points.
quickDASH score | 6 weeks post-operatively
  Secondary analysis will look at all longitudinal evaluation time points of quickDASH using a mixed linear regression model to account for correlations across subjects at multiple time points.
quickDASH score | 12 weeks post-operatively
  Secondary analysis will look at all longitudinal evaluation time points of quickDASH using a mixed linear regression model to account for correlations across subjects at multiple time points.
quickDASH | 6 months post-operatively
  Secondary analysis will look at all longitudinal evaluation time points of quickDASH using a mixed linear regression model to account for correlations across subjects at multiple time points.

CONTACTS AND LOCATIONS:
Overall Officials: Akin Cil, MD, Principal Investigator — University of Missouri-Kansas City Department of Orthopaedic Surgery
Locations (1):
- Truman Medical Centers, Kansas City, Missouri, United States

REFERENCES:
- [Background] Neviaser AS, Hannafin JA. Adhesive capsulitis: a review of current treatment. Am J Sports Med. 2010 Nov;38(11):2346-56. doi: 10.1177/0363546509348048. Epub 2010 Jan 28. PMID 20110457
- [Background] Neviaser JS: Adhesive capsulitis of the shoulder. JBJS 1945;27:211-222.
- [Background] Neviaser RJ, Neviaser TJ. The frozen shoulder. Diagnosis and management. Clin Orthop Relat Res. 1987 Oct;(223):59-64. PMID 3652593
- [Background] Emig EW, Schweitzer ME, Karasick D, Lubowitz J. Adhesive capsulitis of the shoulder: MR diagnosis. AJR Am J Roentgenol. 1995 Jun;164(6):1457-9. doi: 10.2214/ajr.164.6.7754892.
- [Background] Sofka CM, Ciavarra GA, Hannafin JA, Cordasco FA, Potter HG. Magnetic resonance imaging of adhesive capsulitis: correlation with clinical staging. HSS J. 2008 Sep;4(2):164-9. doi: 10.1007/s11420-008-9088-1. Epub 2008 Aug 20. PMID 18815860
- [Background] Miller MD, Wirth MA, Rockwood CA Jr. Thawing the frozen shoulder: the "patient" patient. Orthopedics. 1996 Oct;19(10):849-53. doi: 10.3928/0147-7447-19961001-06. PMID 8905857
- [Background] Griggs SM, Ahn A, Green A. Idiopathic adhesive capsulitis. A prospective functional outcome study of nonoperative treatment. J Bone Joint Surg Am. 2000 Oct;82(10):1398-407. PMID 11057467
- [Background] Shaffer B, Tibone JE, Kerlan RK. Frozen shoulder. A long-term follow-up. J Bone Joint Surg Am. 1992 Jun;74(5):738-46. PMID 1624489
- [Background] Levine WN, Kashyap CP, Bak SF, Ahmad CS, Blaine TA, Bigliani LU. Nonoperative management of idiopathic adhesive capsulitis. J Shoulder Elbow Surg. 2007 Sep-Oct;16(5):569-73. doi: 10.1016/j.jse.2006.12.007. Epub 2007 May 24. PMID 17531513
- [Background] Jones DS, Chattopadhyay C. Suprascapular nerve block for the treatment of frozen shoulder in primary care: a randomized trial. Br J Gen Pract. 1999 Jan;49(438):39-41. PMID 10622015
- [Background] Dodenhoff RM, Levy O, Wilson A, Copeland SA. Manipulation under anesthesia for primary frozen shoulder: effect on early recovery and return to activity. J Shoulder Elbow Surg. 2000 Jan-Feb;9(1):23-6. doi: 10.1016/s1058-2746(00)90005-3. PMID 10717858
- [Background] Farrell CM, Sperling JW, Cofield RH. Manipulation for frozen shoulder: long-term results. J Shoulder Elbow Surg. 2005 Sep-Oct;14(5):480-4. doi: 10.1016/j.jse.2005.02.012. PMID 16194738
- [Background] Ogilvie-Harris DJ, Biggs DJ, Fitsialos DP, MacKay M. The resistant frozen shoulder. Manipulation versus arthroscopic release. Clin Orthop Relat Res. 1995 Oct;(319):238-48. PMID 7554636
- [Background] Pollock RG, Duralde XA, Flatow EL, Bigliani LU. The use of arthroscopy in the treatment of resistant frozen shoulder. Clin Orthop Relat Res. 1994 Jul;(304):30-6. PMID 8020231
- [Background] Warner JJ, Allen AA, Marks PH, Wong P. Arthroscopic release of postoperative capsular contracture of the shoulder. J Bone Joint Surg Am. 1997 Aug;79(8):1151-8. doi: 10.2106/00004623-199708000-00006. PMID 9278074
- [Background] Ozbaydar MU, Tonbul M, Altun M, Yalaman O. [Arthroscopic selective capsular release in the treatment of frozen shoulder]. Acta Orthop Traumatol Turc. 2005;39(2):104-13. Turkish. PMID 15925932
- [Background] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Background] Williams GN, Gangel TJ, Arciero RA, Uhorchak JM, Taylor DC. Comparison of the Single Assessment Numeric Evaluation method and two shoulder rating scales. Outcomes measures after shoulder surgery. Am J Sports Med. 1999 Mar-Apr;27(2):214-21. doi: 10.1177/03635465990270021701. PMID 10102104
- [Background] Hayes K, Walton JR, Szomor ZR, Murrell GA. Reliability of five methods for assessing shoulder range of motion. Aust J Physiother. 2001;47(4):289-94. doi: 10.1016/s0004-9514(14)60274-9. PMID 11722295
- [Background] Hsu JE, Anakwenze OA, Warrender WJ, Abboud JA. Current review of adhesive capsulitis. J Shoulder Elbow Surg. 2011 Apr;20(3):502-14. doi: 10.1016/j.jse.2010.08.023. Epub 2010 Dec 16. No abstract available. PMID 21167743
- [Background] Neviaser AS, Neviaser RJ. Adhesive capsulitis of the shoulder. J Am Acad Orthop Surg. 2011 Sep;19(9):536-42. doi: 10.5435/00124635-201109000-00004. PMID 21885699
- [Background] Vickers AJ. How to randomize. J Soc Integr Oncol. 2006 Fall;4(4):194-8. doi: 10.2310/7200.2006.023. PMID 17022927
- [Background] Campbell MK, Entwistle VA, Cuthbertson BH, Skea ZC, Sutherland AG, McDonald AM, Norrie JD, Carlson RV, Bridgman S; KORAL study group. Developing a placebo-controlled trial in surgery: issues of design, acceptability and feasibility. Trials. 2011 Feb 21;12:50. doi: 10.1186/1745-6215-12-50. PMID 21338481
- [Background] Dempsey AL, Mills T, Karsch RM, Branch TP. Maximizing total end range time is safe and effective for the conservative treatment of frozen shoulder patients. Am J Phys Med Rehabil. 2011 Sep;90(9):738-45. doi: 10.1097/PHM.0b013e318214ed0d. PMID 21430510
- [Background] Angst F, Schwyzer HK, Aeschlimann A, Simmen BR, Goldhahn J. Measures of adult shoulder function: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) and its short version (QuickDASH), Shoulder Pain and Disability Index (SPADI), American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form, Constant (Murley) Score (CS), Simple Shoulder Test (SST), Oxford Shoulder Score (OSS), Shoulder Disability Questionnaire (SDQ), and Western Ontario Shoulder Instability Index (WOSI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S174-88. doi: 10.1002/acr.20630. No abstract available. PMID 22588743
- [Background] Wright RW, Baumgarten KM. Shoulder outcomes measures. J Am Acad Orthop Surg. 2010 Jul;18(7):436-44. doi: 10.5435/00124635-201007000-00006. PMID 20595136